CLINICAL TRIAL: NCT00250276
Title: Assess Lot-to-lot Consistency of GSK Biologicals' HPV-16/18 L1/AS04 Vaccine Following Manufacturing Adjustments Administered Intramuscularly According to a 0,1,6-mth Schedule in Healthy Female Subjects (18-25 y)
Brief Title: Evaluation of the Immune Responses of GSK Biologicals' HPV Vaccine Following Manufacturing Process Adaptation.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 104772; 2005-001667-58 (EudraCT Number)
Record Dates: First submitted 2005-11-07; First posted 2005-11-08 (Estimated); Results first posted 2017-03-17 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Infections, Papillomavirus; Papillomavirus Vaccines
MeSH Terms: conditions — Papillomavirus Infections | interventions — human papillomavirus vaccine, L1 type 16, 18

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Cervarix Lot1 Group (Experimental): Subjects aged between and including 18-25 years, who received one dose of Cervarix™ vaccine Lot 1 manufactured at 600L scale according to a 0, 1, 6- month schedule and were followed up for 7 months after the first dose. Additionally, a telephone contact was foreseen at Month 12. The vaccine was administrated by intramuscular (IM) injection into the deltoid region of the non-dominant arm.
  Interventions: Biological: Cervarix™
- Cervarix Lot2 Group (Experimental): Subjects aged between and including 18-25 years, who received one dose of Cervarix™ vaccine Lot 2 manufactured at 600L scale according to a 0, 1, 6- month schedule and were followed up for 7 months after the first dose. Additionally, a telephone contact was foreseen at Month 12. The vaccine was administrated by intramuscular (IM) injection into the deltoid region of the non-dominant arm.
  Interventions: Biological: Cervarix™
- Cervarix Lot3 Group (Experimental): Subjects aged between and including 18-25 years, who received one dose of Cervarix™ vaccine Lot 3 manufactured at 600L scale according to a 0, 1, 6- month schedule and were followed up for 7 months after the first dose. Additionally, a telephone contact was foreseen at Month 12. The vaccine was administrated by intramuscular (IM) injection into the deltoid region of the non-dominant arm.
  Interventions: Biological: Cervarix™
- Cervarix Low Group (Experimental): Subjects aged between and including 18-25 years, who received one dose of Cervarix™ vaccine manufactured lower scale-80L according to a 0, 1, 6- month schedule and were followed up for 7 months after the first dose. Additionally, a telephone contact was foreseen at Month 12. The vaccine was administrated by intramuscular (IM) injection into the deltoid region of the non-dominant arm.
  Interventions: Biological: Cervarix™

INTERVENTIONS:
Biological: Cervarix™ — GSK Biologicals' vaccine against human papillomaviruses 16 and 18.

SUMMARY:
Human papillomavirus infection has clearly been recognized as the cause of cervical cancer. Indeed, the infection of the cervix by certain oncogenic types of HPV, if not cleared , can lead over time to cervical cancer in women . This study will compare the immune response induced by different lots of the HPV-16/18 L1/AS04 vaccine, following adjustments to the manufacturing process.

ELIGIBILITY:
Inclusion Criteria:

* A female subject between, and including, 18 and 25 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject prior to enrolment.
* Subject must have a negative urine pregnancy test.
* Healthy subject before entering the study entry as established by medical history and physical examination.
* Subject must be of non-childbearing potential.

Exclusion Criteria:

* pregnant or breastfeeding subject.
* previous vaccination against human papillomavirus (HPV).
* Known acute or chronic, clinically significant neurologic, hepatic or renal functional abnormality.
* History of chronic condition(s) requiring treatment such as cancer, chronic hepatic or kidney disease(s), diabetes or autoimmune disease.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 798 (Actual)
Dates: Start 2005-10-28 (Actual); Primary Completion 2007-03-01 (Actual); Study Completion 2007-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- GSK Investigational Site, Hvidovre, Denmark
- Lithuania (3):
  - GSK Investigational Site, Kaunas
  - GSK Investigational Site, Klaipėda
  - GSK Investigational Site, Vilnius
- Poland (3):
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=1515

REFERENCES:
- [Background] Descamps D, Hardt K, Spiessens B, Izurieta P, Verstraeten T, Breuer T, Dubin G. Safety of human papillomavirus (HPV)-16/18 AS04-adjuvanted vaccine for cervical cancer prevention: a pooled analysis of 11 clinical trials. Hum Vaccin. 2009 May;5(5):332-40. doi: 10.4161/hv.5.5.7211. Epub 2009 May 20. PMID 19221517
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 104772 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104772 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 104772 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104772 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104772 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104772 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104772 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cervarix Lot1 Group | Cervarix Lot2 Group | Cervarix Lot3 Group | Cervarix Low Group
Started | 199 | 198 | 201 | 200
Completed | 182 | 177 | 182 | 181
Not Completed | 17 | 21 | 19 | 19
Not completed — Serious Adverse Event | 0 | 0 | 1 | 0
Not completed — Non-serious Adverse Event | 2 | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 3 | 2
Not completed — Migrated/moved from study area | 3 | 0 | 2 | 7
Not completed — Lost to Follow-up | 11 | 18 | 13 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix Lot1 Group | Cervarix Lot2 Group | Cervarix Lot3 Group | Cervarix Low Group | Total
Number analyzed (Participants) | 199 | 198 | 201 | 200 | 798
Age, Continuous [Mean (Standard Deviation); unit: Years] | 21.8 (2.08) | 21.8 (2.08) | 21.9 (2.00) | 22.0 (1.96) | 21.88 (2.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 199 | 198 | 201 | 200 | 798
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted (SCR) Subjects for Anti-Human Papillomavirus Type 16 (Anti-HPV-16) and Anti-Human Papillomavirus Type 18 (Anti-HPV-18)
Description: Seroconversion was defined as the appearance of anti-HPV-16 and/or anti-HPV-18 antibodies (anti-HPV-16 concentrations ≥8 Enzyme-Linked Immunosorbent Assay [ELISA] units per milliliter [EL.U/mL] and anti-HPV-18 concentrations ≥7 EL.U/mL) in the serum of subjects seronegative before vaccination.
Time Frame: At Month 7
Population: The According-to-Protocol cohort for immunogenicity included all evaluable subjects from whom data concerning immunogenicity measures were available. This included subjects for whom assay results were available for antibodies against at least one study vaccine component at Month 7.
Measure: Count of Participants; unit: Participants
Groups:
- Pooled Group: The 3 study groups receiving the 3 different lots of Cervarix™ vaccine manufactured at 600L scale were pooled to demonstrate consistency for data analysis.
Arm/Group | Cervarix Lot1 Group | Cervarix Lot2 Group | Cervarix Lot3 Group | Pooled Group | Cervarix Low Group
Number analyzed (Participants) | 129 | 143 | 135 | 407 | 117
Participants
  Anti-HPV-16: number analyzed (Participants) | 118 | 127 | 126 | 371 | 102
  Anti-HPV-16 | 118 | 127 | 126 | 371 | 102
  Anti-HPV-18 | 129 | 143 | 135 | 407 | 117
Statistical Analysis 1: Comparison: Cervarix Lot1 Group vs Cervarix Lot2 Group; To demonstrate lot-to-lot consistency in terms of immunogenicity between the 3 industrial production lots (600L scale) of the Cervarix™ vaccine, one month post dose 3 (Month 7). If consistency was demonstrated the 3 lots would be pooled and non-inferiority of the 600L scale lot vaccine versus the 80L scale would be evaluated as a second primary objective; Test type: Non-Inferiority or Equivalence — The first primary objective was reached as the 95% Confidence Interval (CI) of the GMC ratio between lots was within [0.5;2] for the anti-HPV-16 antibodies; ANOVA; The ANOVA model on the logarithm (log)10 transformation of the concentrations. The ANOVA model included the vaccine group as fixed effect; GMC ratio for anti-HPV-16 antibody = 1.04, 95% CI 2-sided [0.81 to 1.34]
Statistical Analysis 2: Comparison: Cervarix Lot1 Group vs Cervarix Lot2 Group; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — The first primary objective was reached as the 95% CIs of the GMC ratio between lots were within [0.5;2] for the anti-HPV-18 antibodies; ANOVA; The ANOVA model on the log10 transformation of theconcentrations. The ANOVA model included the vaccine group as fixed effect; GMC ratio for anti-HPV-18 antibody = 1.19, 95% CI 2-sided [0.95 to 1.49]
Statistical Analysis 3: Comparison: Cervarix Lot1 Group vs Cervarix Lot3 Group; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — The first primary objective was reached as the 95% CIs of the GMC ratio between lots were within [0.5;2] for the anti-HPV-16 antibodies; ANOVA; The ANOVA model on the log10 transformation of the concnetration. The ANOVA model included the vaccine group as fixed effect; GMC ratio for anti-HPV-16 antibody = 1.26, 95% CI 2-sided [0.98 to 1.63]
Statistical Analysis 4: Comparison: Cervarix Lot1 Group vs Cervarix Lot3 Group; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; ANOVA; [statistical method as in outcome 1, analysis 3]; GMC ratio for anti-HPV-18 antibody = 1.48, 95% CI 2-sided [1.18 to 1.85]
Statistical Analysis 5: Comparison: Cervarix Lot2 Group vs Cervarix Lot3 Group; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 3]; ANOVA; The ANOVA model on the log10 transformation of the concentration. The ANOVA model included the vaccine group as fixed effect; GMT ratio for anti-HPV-16 antibody = 1.21, 95% CI 2-sided [0.94 to 1.55]
Statistical Analysis 6: Comparison: Cervarix Lot2 Group vs Cervarix Lot3 Group; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; ANOVA; [statistical method as in outcome 1, analysis 5]; GMC ratio for anti-HPV-18 antibody = 1.24, 95% CI 2-sided [1.00 to 1.55]
Statistical Analysis 7: Comparison: Pooled Group vs Cervarix Low Group; To demonstrate that the Cervarix™ vaccine produced at 600L manufacturing scale was non-inferior in terms of immunogenicity to the Cervarix™ vaccine produced at 80L scale, one month after the third dose (Month 7); Test type: Non-Inferiority or Equivalence — The second primary objective was reached as the upper limit of the 95% CI of the difference in seroconversion rates for anti-HPV-16 antibodies was below 5%; Proc StatXact 5.0; Difference in seroconversion rate = 0.00, 95% CI 2-sided [-3.63 to 1.02]
Statistical Analysis 8: Comparison: Pooled Group vs Cervarix Low Group; To demonstrate that the Cervarix™ vaccine produced at 600L manufacturing scale was non-inferior in terms of immunogenicity to the Cervarix™ vaccine produced at 80L scale, on month after the third dose (Month 7); Test type: Non-Inferiority or Equivalence — The second primary objective was reached as the upper limit of the 95% CI of the difference in seroconversion rates for anti-HPV-18 antibodies was below 5%; Proc StatXact 5.0; Difference in seroconversion rate = 0.00, 95% CI 2-sided [-3.18 to 0.94]
Statistical Analysis 9: Comparison: Pooled Group vs Cervarix Low Group; [analysis description as in outcome 1, analysis 8]; Test type: Non-Inferiority or Equivalence — The second primary objective was reached as the upper limit of the 95% CI of the GMC rates for anti-HPV-16 was below 2%; ANOVA; The ANOVA model on the log10 transformation of the concentration, included the vaccine groups as fixed effect (pooled 600L lot versus 80L lot); GMC ratio for anti-HPV-16 antibody = 0.87, 95% CI 2-sided [0.70 to 1.08]
Statistical Analysis 10: Comparison: Pooled Group vs Cervarix Low Group; [analysis description as in outcome 1, analysis 8]; Test type: Non-Inferiority or Equivalence — The second primary objective was reached as the upper limit of the 95% CI of the GMC rates anti-HPV-18 antibodies was below 2%; ANOVA; [statistical method as in outcome 1, analysis 9]; GMC ratio for anti-HPV-18 antibody = 0.80, 95% CI 2-sided [0.66 to 0.97]

2. Primary Outcome: Number of Seropositive Subjects for Anti-HPV-16 and Anti-HPV-18
Description: Seropositivity defined subjects with anti-HPV-16 antibody concentration ≥ 8 EL.U/mL and/or anti-HPV-18 antibody concentration ≥ 7 EL.U/mL.
Time Frame: At Month 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Lot1 Group | Cervarix Lot2 Group | Cervarix Lot3 Group | Cervarix Low Group
Number analyzed (Participants) | 54 | 38 | 43 | 57
Participants
  Anti-HPV-16 | 54 | 38 | 43 | 57
  Anti-HPV-18: number analyzed (Participants) | 43 | 22 | 34 | 41
  Anti-HPV-18 | 43 | 22 | 34 | 41

3. Secondary Outcome: Number of SCR Subjects for Anti-HPV-16 and Anti-HPV-18
Description: Seroconversion was defined as the appearance of anti-HPV-16 and/or anti-HPV-18 antibodies (anti-HPV-16 concentrations ≥8 ELISA units per milliliter [EL.U/mL] and anti-HPV-18 concentrations ≥7 EL.U/mL) in the serum of subjects seronegative before vaccination.
Time Frame: At Month 2
Population: The According-to-Protocol cohort for immunogenicity included all evaluable subjects from whom data concerning immunogenicity measures were available. This included subjects for whom assay results were available for antibodies against at least one study vaccine component at Month 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Lot1 Group | Cervarix Lot2 Group | Cervarix Lot3 Group | Cervarix Low Group
Number analyzed (Participants) | 128 | 142 | 134 | 116
Participants
  Anti-HPV-16: number analyzed (Participants) | 117 | 126 | 125 | 102
  Anti-HPV-16 | 117 | 126 | 125 | 102
  Anti-HPV-18 | 128 | 142 | 134 | 116

4. Secondary Outcome: Number of Seropositive Subjects for Anti-HPV-16 and Anti-HPV-18
Description: Seropositivity defined subjects with anti-HPV-16 antibody concentration ≥ 8 EL.U/mL and/or anti-HPV-18 antibody concentration ≥ 7 EL.U/mL .
Time Frame: At Month 2
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Lot1 Group | Cervarix Lot2 Group | Cervarix Lot3 Group | Cervarix Low Group
Number analyzed (Participants) | 54 | 38 | 43 | 56
Participants
  Anti-HPV-16 | 54 | 38 | 43 | 56
  Anti-HPV-18: number analyzed (Participants) | 43 | 22 | 34 | 41
  Anti-HPV-18 | 43 | 22 | 34 | 41

5. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) diameter of injection site.
Time Frame: During the 7-days (Day 0-6) post-vaccination
Population: The Total Vaccinated cohort included all vaccinated subjects. The Total vaccinated cohort for analysis of safety included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Lot1 Group | Cervarix Lot2 Group | Cervarix Lot3 Group | Pooled Group | Cervarix Low Group
Number analyzed (Participants) | 198 | 197 | 199 | 594 | 197
Participants
  Any Pain Dose 1: number analyzed (Participants) | 198 | 197 | 199 | 594 | 196
  Any Pain Dose 1 | 188 | 190 | 178 | 556 | 185
  Grade 3 Pain Dose 1: number analyzed (Participants) | 198 | 197 | 199 | 594 | 196
  Grade 3 Pain Dose 1 | 20 | 16 | 17 | 53 | 12
  Any Redness Dose 1: number analyzed (Participants) | 198 | 197 | 199 | 594 | 196
  Any Redness Dose 1 | 74 | 71 | 77 | 222 | 75
  Grade 3 Redness Dose 1: number analyzed (Participants) | 198 | 197 | 199 | 594 | 196
  Grade 3 Redness Dose 1 | 0 | 0 | 0 | 0 | 0
  Any Swelling Dose 1: number analyzed (Participants) | 198 | 197 | 199 | 594 | 196
  Any Swelling Dose 1 | 58 | 57 | 57 | 172 | 54
  Grade 3 Swelling Dose 1: number analyzed (Participants) | 198 | 197 | 199 | 594 | 196
  Grade 3 Swelling Dose 1 | 9 | 2 | 2 | 13 | 4
  Any Pain Dose 2: number analyzed (Participants) | 196 | 195 | 198 | 589 | 194
  Any Pain Dose 2 | 167 | 166 | 170 | 503 | 161
  Grade 3 Pain Dose 2: number analyzed (Participants) | 196 | 195 | 198 | 589 | 194
  Grade 3 Pain Dose 2 | 17 | 10 | 19 | 46 | 12
  Any Redness Dose 2: number analyzed (Participants) | 196 | 195 | 198 | 589 | 194
  Any Redness Dose 2 | 78 | 85 | 79 | 242 | 62
  Grade 3 Redness Dose 2: number analyzed (Participants) | 196 | 195 | 198 | 589 | 194
  Grade 3 Redness Dose 2 | 3 | 6 | 0 | 9 | 1
  Any Swelling Dose 2: number analyzed (Participants) | 196 | 195 | 198 | 589 | 194
  Any Swelling Dose 2 | 64 | 59 | 56 | 179 | 53
  Grade 3 Swelling Dose 2: number analyzed (Participants) | 196 | 195 | 198 | 589 | 194
  Grade 3 Swelling Dose 2 | 7 | 2 | 2 | 11 | 5
  Any Pain Dose 3: number analyzed (Participants) | 181 | 178 | 184 | 543 | 181
  Any Pain Dose 3 | 164 | 151 | 162 | 477 | 156
  Grade 3 Pain Dose 3: number analyzed (Participants) | 181 | 178 | 184 | 543 | 181
  Grade 3 Pain Dose 3 | 21 | 14 | 11 | 46 | 15
  Any Redness Dose 3: number analyzed (Participants) | 181 | 178 | 184 | 543 | 181
  Any Redness Dose 3 | 94 | 102 | 96 | 292 | 92
  Grade 3 Redness Dose 3: number analyzed (Participants) | 181 | 178 | 184 | 543 | 181
  Grade 3 Redness Dose 3 | 5 | 6 | 4 | 15 | 5
  Any Swelling Dose 3: number analyzed (Participants) | 181 | 178 | 184 | 543 | 181
  Any Swelling Dose 3 | 92 | 84 | 85 | 261 | 82
  Grade 3 Swelling Dose 3: number analyzed (Participants) | 181 | 178 | 184 | 543 | 181
  Grade 3 Swelling Dose 3 | 8 | 3 | 2 | 13 | 3
  Any Pain Across | 194 | 192 | 190 | 576 | 192
  Grade 3 Pain Across | 45 | 29 | 34 | 108 | 30
  Any Redness Across | 118 | 128 | 127 | 373 | 126
  Grade 3 Redness Across | 8 | 9 | 4 | 21 | 6
  Any Swelling Across | 116 | 112 | 113 | 341 | 107
  Grade 3 Swelling Across | 15 | 6 | 6 | 27 | 10

6. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were arthralgia, fatigue, fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)], gastro-intestinal, headache, myalgia, rash and urticaria. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination. Arthralgia (joint pain) = pain occurring in joints that were distal from the injection site. This outcome presents solicited general symptoms post dose 1 of vaccination.
Time Frame: During the 7-days (Day 0-6) post-vaccination
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Lot1 Group | Cervarix Lot2 Group | Cervarix Lot3 Group | Pooled Group | Cervarix Low Group
Number analyzed (Participants) | 198 | 197 | 199 | 594 | 196
Participants
  Any Arthralgia | 19 | 19 | 13 | 51 | 17
  Grade 3 Arthralgia | 1 | 0 | 2 | 3 | 0
  Related Arthralgia | 14 | 17 | 8 | 39 | 14
  Any Fatigue | 81 | 84 | 73 | 238 | 80
  Grade 3 Fatigue | 4 | 1 | 4 | 9 | 5
  Related Fatigue | 60 | 62 | 48 | 170 | 61
  Any Fever | 4 | 7 | 4 | 15 | 5
  Grade 3 Fever | 0 | 0 | 0 | 0 | 0
  Related Fever | 1 | 5 | 3 | 9 | 3
  Any Gastro-intestinal | 32 | 39 | 34 | 105 | 30
  Grade 3 Gastro-intestinal | 1 | 2 | 0 | 3 | 1
  Related Gastro-intestinal | 17 | 24 | 19 | 60 | 19
  Any Headache | 69 | 70 | 60 | 199 | 65
  Grade 3 Headache | 8 | 4 | 2 | 14 | 4
  Related Headache | 44 | 49 | 38 | 131 | 46
  Any Myalgia | 45 | 55 | 50 | 150 | 42
  Grade 3 Myalgia | 3 | 2 | 3 | 8 | 0
  Related Myalgia | 36 | 44 | 41 | 121 | 30
  Any Rash | 4 | 4 | 6 | 14 | 5
  Grade 3 Rash | 0 | 0 | 0 | 0 | 0
  Related Rash | 2 | 3 | 4 | 9 | 4
  Any Urticaria | 5 | 3 | 3 | 11 | 4
  Grade 3 Urticaria | 0 | 0 | 0 | 0 | 0
  Related Urticaria | 2 | 2 | 2 | 6 | 4

7. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were arthralgia, fatigue, fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)], gastro-intestinal, headache, myalgia, rash and urticaria. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination. Arthralgia (joint pain) = pain occurring in joints that were distal from the injection site. This outcome presents solicited general symptoms post dose 2 of vaccination.
Time Frame: During the 7-days (Day 0-6) post-vaccination
Population: The Total Vaccinated cohort included all vaccinated subjects. The Total vaccinated cohort for analysis of safety included all subjects with at last one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Lot1 Group | Cervarix Lot2 Group | Cervarix Lot3 Group | Pooled Group | Cervarix Low Group
Number analyzed (Participants) | 195 | 195 | 198 | 588 | 193
Participants
  Any Arthralgia | 14 | 14 | 14 | 42 | 17
  Grade 3 Arthralgia | 0 | 0 | 1 | 1 | 0
  Related Arthralgia | 12 | 11 | 10 | 33 | 14
  Any Fatigue | 63 | 73 | 69 | 205 | 58
  Grade 3 Fatigue | 2 | 4 | 3 | 9 | 5
  Related Fatigue | 39 | 55 | 38 | 132 | 40
  Any Fever | 7 | 5 | 7 | 19 | 5
  Grade 3 Fever | 0 | 0 | 0 | 0 | 0
  Related Fever | 5 | 2 | 2 | 9 | 3
  Any Gastro-intestinal | 22 | 21 | 28 | 71 | 24
  Grade 3 Gastro-intestinal | 1 | 0 | 1 | 2 | 1
  Related Gastro-intestinal | 14 | 14 | 12 | 40 | 9
  Any Headache | 47 | 51 | 46 | 144 | 41
  Grade 3 Headache | 2 | 4 | 2 | 8 | 1
  Related Headache | 27 | 33 | 29 | 89 | 24
  Any Myalgia | 30 | 37 | 39 | 106 | 31
  Grade 3 Myalgia | 0 | 1 | 3 | 4 | 1
  Related Myalgia | 22 | 30 | 31 | 83 | 21
  Any Rash | 1 | 3 | 8 | 12 | 5
  Grade 3 Rash | 0 | 0 | 0 | 0 | 0
  Related Rash | 1 | 3 | 5 | 9 | 3
  Any Urticaria | 2 | 2 | 2 | 6 | 5
  Grade 3 Urticaria | 0 | 0 | 0 | 0 | 0
  Related Urticaria | 0 | 1 | 2 | 3 | 3

8. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were arthralgia, fatigue, fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)], gastro-intestinal, headache, myalgia, rash and urticaria. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination. Arthralgia (joint pain) = pain occurring in joints that were distal from the injection site. This outcome presents solicited general symptoms post dose 3 of vaccination.
Time Frame: During the 7-days (Day 0-6) post-vaccination
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Lot1 Group | Cervarix Lot2 Group | Cervarix Lot3 Group | Pooled Group | Cervarix Low Group
Number analyzed (Participants) | 181 | 178 | 184 | 543 | 181
Participants
  Any Arthralgia | 18 | 19 | 18 | 55 | 13
  Grade 3 Arthralgia | 1 | 1 | 0 | 2 | 0
  Related Arthralgia | 15 | 16 | 12 | 43 | 11
  Any Fatigue | 76 | 67 | 64 | 207 | 60
  Grade 3 Fatigue | 9 | 1 | 2 | 12 | 6
  Related Fatigue | 58 | 50 | 49 | 157 | 49
  Any Fever | 7 | 6 | 4 | 17 | 8
  Grade 3 Fever | 0 | 0 | 1 | 1 | 0
  Related Fever | 1 | 4 | 1 | 6 | 4
  Any Gastro-intestinal | 17 | 19 | 25 | 61 | 15
  Grade 3 Gastro-intestinal | 2 | 1 | 1 | 4 | 3
  Related Gastro-intestinal | 8 | 9 | 14 | 31 | 7
  Any Headache | 53 | 44 | 49 | 146 | 39
  Grade 3 Headache | 5 | 2 | 4 | 11 | 1
  Related Headache | 34 | 31 | 29 | 94 | 30
  Any Myalgia | 44 | 38 | 39 | 121 | 29
  Grade 3 Myalgia | 3 | 2 | 1 | 6 | 1
  Related Myalgia | 35 | 35 | 32 | 102 | 24
  Any Rash | 7 | 4 | 9 | 20 | 9
  Grade 3 Rash | 0 | 0 | 0 | 0 | 0
  Related Rash | 5 | 2 | 6 | 13 | 6
  Any Urticaria | 3 | 0 | 5 | 8 | 6
  Grade 3 Urticaria | 0 | 0 | 0 | 0 | 0
  Related Urticaria | 1 | 0 | 2 | 3 | 4

9. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were arthralgia, fatigue, fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)], gastro-intestinal, headache, myalgia, rash and urticaria. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination. Arthralgia (joint pain) = pain occurring in joints that were distal from the injection site. This outcome presents results across vaccination doses for solicited general symptoms.
Time Frame: During the 7-days (Day 0-6) post-vaccination
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Lot1 Group | Cervarix Lot2 Group | Cervarix Lot3 Group | Pooled Group | Cervarix Low Group
Number analyzed (Participants) | 198 | 197 | 199 | 594 | 197
Participants
  Any Arthralgia | 38 | 40 | 32 | 110 | 35
  Grade 3 Arthralgia | 2 | 1 | 2 | 5 | 0
  Related Arthralgia | 31 | 32 | 22 | 85 | 31
  Any Fatigue | 117 | 117 | 106 | 340 | 105
  Grade 3 Fatigue | 13 | 6 | 8 | 27 | 12
  Related Fatigue | 90 | 95 | 78 | 263 | 90
  Any Fever | 16 | 18 | 14 | 48 | 15
  Grade 3 Fever | 0 | 0 | 1 | 1 | 0
  Related Fever | 6 | 11 | 5 | 22 | 7
  Any Gastro-intestinal | 55 | 61 | 57 | 173 | 49
  Grade 3 Gastro-intestinal | 4 | 3 | 2 | 9 | 5
  Related Gastro-intestinal | 32 | 38 | 33 | 103 | 25
  Any Headache | 99 | 103 | 95 | 297 | 93
  Grade 3 Headache | 14 | 9 | 8 | 31 | 5
  Related Headache | 68 | 77 | 57 | 202 | 68
  Any Myalgia | 75 | 82 | 73 | 230 | 66
  Grade 3 Myalgia | 6 | 5 | 6 | 17 | 2
  Related Myalgia | 62 | 70 | 62 | 194 | 48
  Any Rash | 11 | 10 | 19 | 40 | 15
  Grade 3 Rash | 0 | 0 | 0 | 0 | 0
  Related Rash | 7 | 7 | 13 | 27 | 11
  Any Urticaria | 7 | 5 | 7 | 19 | 10
  Grade 3 Urticaria | 0 | 0 | 0 | 0 | 0
  Related Urticaria | 3 | 3 | 4 | 10 | 8

10. Secondary Outcome: Number of Subjects With New Onset Chronic Diseases (NOCDs)
Description: NOCDs include autoimmune disorders, asthma, type I diabetes, allergies.
Time Frame: From Month 0 to Month 7
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Lot1 Group | Cervarix Lot2 Group | Cervarix Lot3 Group | Pooled Group | Cervarix Low Group
Number analyzed (Participants) | 199 | 198 | 201 | 598 | 200
Participants | 3 | 4 | 7 | 14 | 3

11. Secondary Outcome: Number of Subjects With Medically Significant Adverse Events (MSAEs)
Description: MSAEs prompting emergency room or physician visits that are not related to common diseases or routine visits for physical examination or vaccination, or serious adverse events (SAEs) that are not related to common diseases. Common diseases include upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervico-vaginal yeast infections, menstrual cycle abnormalities and injury.
Time Frame: From Month 0 to Month 7
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Groups:
- Cervarix Low Group: Subjects aged between and including 18-25 years, who received one dose of Cervarix™ vaccine manufactured at lower scale-80L according to a 0, 1, 6- month schedule and were followed up for 7 months after the first dose. Additionally, a telephone contact was foreseen at Month 12. The vaccine was administrated by intramuscular (IM) injection into the deltoid region of the non-dominant arm.
Arm/Group | Pooled Group | Cervarix Low Group
Number analyzed (Participants) | 598 | 200
Participants | 71 | 23

12. Secondary Outcome: Number of Subjects With (NOCDs)
Description: NOCDs include autoimmune disorders, asthma, type I diabetes, allergies.
Time Frame: From Month 0 to Month 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Lot1 Group | Cervarix Lot2 Group | Cervarix Lot3 Group | Pooled Group | Cervarix Low Group
Number analyzed (Participants) | 199 | 198 | 201 | 598 | 200
Participants | 4 | 4 | 7 | 15 | 3

13. Secondary Outcome: Number of Subjects With MSAEs
Description: as for outcome 11
Time Frame: From Month 0 to Month 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Group | Cervarix Low Group
Number analyzed (Participants) | 598 | 200
Participants | 78 | 23

14. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: Within 30 days (Day 0-29) post vaccination
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Lot1 Group | Cervarix Lot2 Group | Cervarix Lot3 Group | Pooled Group | Cervarix Low Group
Number analyzed (Participants) | 199 | 198 | 201 | 598 | 200
Participants
  Any (AEs) | 58 | 56 | 76 | 190 | 67
  Grade 3 (AEs) | 5 | 6 | 14 | 25 | 7
  Related (AEs) | 22 | 23 | 30 | 75 | 32

15. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Month 0 to Month 7
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Lot1 Group | Cervarix Lot2 Group | Cervarix Lot3 Group | Pooled Group | Cervarix Low Group
Number analyzed (Participants) | 199 | 198 | 201 | 598 | 200
Participants | 2 | 0 | 2 | 4 | 3

16. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 15
Time Frame: From Month 0 to Month 12
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Lot1 Group | Cervarix Lot2 Group | Cervarix Lot3 Group | Pooled Group | Cervarix Low Group
Number analyzed (Participants) | 199 | 198 | 201 | 598 | 200
Participants | 6 | 1 | 2 | 9 | 3

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms: during the 7-days (Day 0-6) post vaccination. AEs: during the 30-days (Day 0-29) post vaccination. SAEs throughout the whole study period (up to Month 12).
Arm/Group | Cervarix Lot1 Group | Cervarix Lot2 Group | Cervarix Lot3 Group | Pooled Group | Cervarix Low Group
Serious Adverse Events (participants affected / at risk) | 6/199 | 1/198 | 2/201 | 9/598 | 3/200
Other Adverse Events (participants affected / at risk) | 196/199 | 194/198 | 191/201 | 581/598 | 194/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Lot1 Group (N=199) | Cervarix Lot2 Group (N=198) | Cervarix Lot3 Group (N=201) | Pooled Group (N=598) | Cervarix Low Group (N=200)
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Basedow's disease (Endocrine disorders) | 1 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Cerebral malaria (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Pelvic inflammatory disease (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4.9% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cervarix Lot1 Group (N=199) | Cervarix Lot2 Group (N=198) | Cervarix Lot3 Group (N=201) | Pooled Group (N=598) | Cervarix Low Group (N=200)
Pain (General disorders) | 194/198 | 192/197 | 190/199 | 576/594 | 192/197
Redness (General disorders) | 118/198 | 128/197 | 127/199 | 373/594 | 126/197
Swelling (General disorders) | 116/198 | 112/197 | 113/199 | 341/594 | 107/197
Arthralgia (General disorders) | 38/198 | 40/197 | 32/199 | 110/594 | 35/197
Fatigue (General disorders) | 117/198 | 117/197 | 106/199 | 340/594 | 105/197
Fever/(Axillary) (°C) (General disorders) | 16/198 | 18/197 | 14/199 | 48/594 | 15/197
Gastrointestinal (General disorders) | 55/198 | 61/197 | 57/199 | 173/594 | 49/197
Headache (General disorders) | 99/198 | 103/197 | 95/199 | 297/594 | 93/197
Myalgia (General disorders) | 75/198 | 82/197 | 73/199 | 230/594 | 66/197
Rash (General disorders) | 11/198 | 10/197 | 19/199 | 40/594 | 15/197
Urticaria (General disorders) | 7/198 | 5/197 | 7/199 | 19/594 | 10/197
Injection site pruritus (General disorders) | 7 | 3 | 4 | 14 | 10
Nasopharyngitis (Infections and infestations) | 8 | 8 | 10 | 26 | 7

LIMITATIONS AND CAVEATS:
None reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.